CLINICAL TRIAL: NCT06154525
Title: Evaluating the Effectiveness of the LiveSpo® Preg-Mom and LiveSpo® KIDS Spore Probiotics in Supporting the Reduction of Constipation, Anorexia, and Slow Weight Gain in Children Aged 24-60 Months
Brief Title: Effectiveness of Bacillus Spore Probiotics in Reducing Constipation, Anorexia, and Slow Weight Gain in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anabio R&D (Industry)
Collaborators: National Institute of Nutrition, Vietnam (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TNLS 2023.1224/QLKH-VDD
Record Dates: First submitted 2023-11-16; First posted 2023-12-04 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Constipation; Anorexia; Weight Gain
Keywords: Bacillus spore; Children; Gut microbiota; Cytokine
MeSH Terms: conditions — Constipation; Anorexia; Weight Gain

STUDY DESIGN:
Intervention Model Description: A randomized, double-blind, controlled clinical trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: LiveSpo Preg - Mom, LiveSpo KIDS, and RO water are indistinguishable regarding smell and taste. Because the three liquid products are packed in opaque plastic ampoules, the color and turbidity of the suspension are unrecognizable to investigators, trainers, the patient's parents, and patients except for the Principal Investigator (PI) and final data analysis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control Group (CC) (Placebo Comparator): The control group receives RO water with a dosage of 1 ampoule per time, 2 times per day for 28 days.
  Interventions: Other: RO water
- Preg-Mom Group (AA) (Experimental): The Preg-Mom group receives RO water plus B. subtilis, B. clausii, and B. coagulans at 3 billion CFU/5 mL (LiveSpo® Preg-Mom) with a dosage of 1 ampoule per time, 2 times per day for 28 days.
  Interventions: Dietary Supplement: LiveSpo Preg-Mom
- KIDS Group (BB) (Experimental): The KIDS group receives RO water plus B. subtilis and B. clausii at 3 billion CFU/5 mL (LiveSpo® KIDS) with a dosage of 1 ampoule per time, 2 times per day for 28 days.
  Interventions: Dietary Supplement: LiveSpo KIDS

INTERVENTIONS:
Other: RO water — Aquafina's reverse osmosis (RO) water, produced by PepsiCo, have both obtained ISO 9001:2015 and ISO 22000:2018 certifications, which are internationally recognized standards for quality management and food safety management systems, respectively. The RO water ampoules are produced using a similar process as the LIVESPO Preg-Mom/ KIDS but contain 5ml of high-quality RO water from Aquafina (proper noun)
  Arms: Control Group (CC)
Dietary Supplement: LiveSpo Preg-Mom — LiveSpo® Preg-Mom has a registration number 7695/2020/ĐKSP issued by the Food Safety Department of the Ministry of Health in Vietnam.
  Arms: Preg-Mom Group (AA)
Dietary Supplement: LiveSpo KIDS — LiveSpo® KIDS has a registration number 1537/2023/ĐKSP issued by the Food Safety Department of the Ministry of Health in Vietnam.
  Arms: KIDS Group (BB)

SUMMARY:
Constipation is rising globally and is a health concern in Asia. Prolonged constipation, without proper care, can lead to complications affecting a child's physical and psychological development, causing significant health and socioeconomic impacts. Anorexia is also common in children, affecting their nutrient absorption, weight gain, and height development. Anorexic children are 2.5-3 times more likely to suffer from underweight and stunting. A number of studies have suggested that probiotics can reduce stool retention time and improve stool consistency, making them a natural and safe option for relieving constipation in adults and children. Probiotics, particularly spore-forming probiotics like Bacillus clausii, Bacillus subtilis, and Bacillus coagulans, have shown promise in improving gut health and combating anorexia, constipation, and malnutrition. With this background, the investigators conduct a research project titled "Evaluating the effectiveness of the LiveSpo® Preg-Mom and LiveSpo® KIDS in supporting the reduction of constipation, anorexia, and slow weight gain in children aged 24-60 months".

The study aims to: (i) Evaluate the effectiveness of LiveSpo® Preg-Mom and LiveSpo® KIDS in reducing constipation, anorexia, and slow weight gain in children. (ii) Assessing the impact of probiotic supplementation on pro-inflammatory/anti-inflammatory cytokines concentrations in the blood, IgA concentrations in stools, and changes in the intestinal microbiota composition in the children's stools.

Study Population: The sample size for aims is 201. Description of Sites: the study is conducted at three communes in Vo Nhai district, Thai Nguyen province.

Description of Study Intervention: 201 eligible children aged 24-60 months with signs of anorexia, constipation, and meeting nutritional criteria were selected. The selected children are randomly assigned to three experiment groups, with 67 children per group. Blood samples are taken (at the start and after 28 days of intervention), and fecal samples are collected at the beginning of the study day, day 7, and day 28 of intervention, to analyze cytokine, IgA concentrations, and the gut microbiota. The intervention products are labeled with three codes corresponding to the three experiment groups (For example AA code is used for LiveSpo® Preg-Mom, BB code for LiveSpo® KIDS, CC for code for RO water) and these codes can be interchanged as needed.

Study duration: 12 months

DETAILED DESCRIPTION:
Child malnutrition is a pressing public health concern, particularly among those under 5 years old, affecting physical, mental, and motor development, leading to chronic issues in adulthood and future generations. A report by UNICEF, WHO, and the World Bank (March 2020) emphasized the alarming global malnutrition rates, with 144.0 million children under 5 experiencing malnutrition, including stunting (47.0 million) and severe malnutrition (14.3 million). Lower-middle-income countries bear the brunt, with two-thirds of stunted and three-quarters of wasted children worldwide. In Vietnam (2020 data), 19.5% of children under 5 are stunted, 11.6% underweight, and 4.7% wasted. In parallel, constipation is a rising health issue in Asia and worldwide, affecting children even in developed economies. Functional constipation is prevalent in children (12-28%). In Vietnam, 24.6% of 3-5-year-olds face constipation, peaking at 54.9% between 36 and 48 months. Untreated constipation poses severe physical, psychological, and socioeconomic complications, such as gastrointestinal inflammation, anorexia, and nutrient malabsorption. Anorexia, prevalent in children, affects their nutrient absorption, growth, and height. Anorexic children have 2.5-3 times higher risks of underweight malnutrition and stunting. Children suffering from malnutrition and digestive disorders face impaired enzyme production, nutrient loss, and gut dysbiosis, causing slow weight gain. Malnourished children with lower immunity become more ill-prone, exacerbating anorexia and forming a problematic cycle. In recent years, the role of probiotics in human health and disease has attracted the attention of researchers. This may be partly due to the excellent activity of probiotics in preventing and alleviating illness. Currently, research on probiotics mainly focuses on treating gastrointestinal diseases with some traditional probiotics. However, a problem arises when adding these microorganisms can hardly survive in extremely harsh environments. Therefore, spore-forming probiotics have attracted the interest of researchers. The viability and stability of these bacteria are significantly better when compared to other probiotics due to their spore-forming ability. Among Bacillus species, Bacillus clausii, Bacillus subtilis, and Bacillus coagulans are bacteria that can form spores stable in the acidic environment of gastric juice and, therefore, pass through the stomach safely and also produce digestive enzymes such as amylase and protease in the intestine. B. coagulans is the only Bacillus species that can produce lactic acid, which reduces the pH, bringing the environment to a slightly acidic status. This is an excellent environmental condition for beneficial intestinal bacteria to grow and prevent the growth of harmful bacteria. At the same time, it enhances absorption and improves anorexia and constipation in children. Previous studies also have demonstrated that probiotics can significantly reduce stool retention time in the intestines and improve stool consistency. Based on the research results above, spore probiotics can be considered natural and safe agents to relieve constipation, anorexia, and slow weight gain in children. To substantiate this argument, the investigators plan to conduct a clinical trial titled "Evaluating the effectiveness of the LiveSpo® Preg-Mom and LiveSpo® KIDS spore probiotics in supporting the reduction of constipation, anorexia, and slow weight gain in children aged 24-60 months".

The overall aim of this study is to assess the efficacy of two types of probiotics, the first one containing 3 billion spores of three bacterial species, Bacillus subtilis, B. clausii, and B. coagulans spores (LiveSpo® Preg-Mom) per ampoule and the second one having 3 billion spores of two bacterial species per ampoule (LiveSpo® KIDS), including Bacillus subtilis, and B. clausii, in supporting the treatment of children with constipation, anorexia, and slow weight gain.

The first objective is to evaluate the effectiveness of these products in alleviating typical symptoms of constipation, anorexia, and slow weight gain. The secondary aim is measuring changes in typical cytokines in the blood, in IgA indices in stool, and microbiota composition in stool before and after supplemental usages of with LiveSpo® Preg-Mom and LiveSpo® KIDS.

For this aim, the study is designed as a randomized, double-blind, and controlled clinical trial with 201 participants diagnosed with constipation, anorexia, and slow weight gain. The participants are randomized into 3 groups using permuted block randomization: a control group using RO water (CC), experimental group 1 using LiveSpo® Preg-Mom (AA), and experimental group 2 using LiveSpo® KIDS (BB). Each patient receives 2 ampoules of the assigned probiotic product daily, divided into 2 doses daily. The study includes clinical assessment of indicators at days 0, 7, and 28, such as weight, types of stool, frequency of daily bowel movements, and average eating time per meal.

Contents and Methods for sub-clinical detection. The study participants are children aged 24 to 60 months who are diagnosed with constipation, anorexia, and slow weight gain.

* Hematology and biochemical tests are conducted on days 0 and 28 at MEDLATEC (proper noun) hospital, Vietnam.
* A real-time PCR assay is conducted on stool samples at days 0, 7, and 28 at the Spobiotic Research Center (proper noun) to detect probiotic spores, including B. subtilis, B. clausii, and B. coagulans, to cross-check the appropriate usage of probiotics or placebo in the experimental and control groups, respectively.
* ELISA tests are conducted at days 0, 7, and 28 at the Spobiotic Research Center (proper noun) to determine pro-inflammatory/ anti-inflammatory cytokine levels in blood samples and IgA levels in stool samples, respectively, for evaluating changes in immune-related indicators during the supportive treatment.
* The tests indicating ratios of bacteria Gr (+) and Gr (-) in stool samples are conducted at days 0, 7, and 28 at MEDLATEC (proper noun) hospital, in order to: evaluate the change in the balance between the types of bacteria Gr (+) and Gr (-) bacteria in gut.
* The 16S V3-V4 metagenome sequencing analysis is carried out at Macrogen (Seoul, Korea) using next-generation sequencing (NGS) technology on the Illumina MiSeq platform (Illumina, San Diego, CA, USA), utilizing a 2 × 250 bp run configuration. DNA samples extracted from stool samples of about 10 representative patients from each group on day 0 and day 28 are used for the analysis, to identify changes in the microbiome.
* Data collection and statistical analysis involve the collection of individual medical records and systematizing patient information into a dataset.

The tabular analysis is performed on dichotomous variables using the χ2 test or Fisher's exact test when the expected value of any cell is below five. Continuous variables are compared using the Wilcoxon test, t-test, or the Mann-Whitney test when data are not normally distributed. To determine if there is a statistically significant difference between the three groups, an ANOVA test is performed. Spearman's correlation analysis assesses the correlations among the variables. Statistical and graphical analyses are performed on GraphPad Prism v8.4.3 software (GraphPad Software, CA, USA). The significance level of all analyses is set at p < 0.05. P-values. The efficacy of LiveSpo® Preg-Mom and LiveSpo® KIDS is evaluated and compared to the control based on the following clinical and sub-clinical criteria obtained from the Experiment and Control groups: Primary outcome is: (i) Symptomatic relief of constipation, anorexia, and slow weight gain; Secondary outcomes are: (ii) Regulated levels of pro-inflammatory cytokines such as IL-6, IL-10, IL-17, IL-23 and TNF-alpha in blood samples. (iii) Regulated IgA levels in fecal samples. (iv) Improved diversity and count of beneficial bacterial species compared to harmful bacteria in the gut microbiota.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 24-60 months.
* Children diagnosed with loss of appetite and/or constipation and/or diarrhea.
* Have a weight-for-age Z-score between -1 and -3.
* Children are fed via the digestive system and have been weaned from breastfeeding.
* The child's parent or guardian agrees to participate in the research and must provide a voluntary commitment letter to comply with the research requirements.

Exclusion Criteria:

* Children outside the age range of 24-60 months
* Severely malnourished children with WAZ-Score > 3, HAZ-Score > 3.
* Currently suffering from acute infectious diseases such as pneumonia, acute diarrhea, liver or kidney disorders, etc.
* Children with a history of preterm birth, low birth weight < 2,500 grams, and twin-twin transfusion syndrome.
* Afflicted with chronic conditions or congenital disabilities, such as Crohn's disease or celiac disease.
* Children using laxatives or other probiotic supplements before the intended research or simultaneously using other probiotics during the research period.
* Parents or guardians who do not consent to participate in the research or do not comply with the research procedures

Ages: 24 Months to 60 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 201 (Actual)
Dates: Start 2024-03-10 (Actual); Primary Completion 2024-04-07 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Changes in the frequency of bowel movements per week | Day 7 compared to Day 0 and Day 28 compared to Day 0
  Changes in the frequency of bowel movements per week (times/week)
Changes in the type of stool based on the Bristol Stool Scale | Day 7 compared to Day 0 and Day 28 compared to Day 0
  Changes in the type of stool based on the Bristol Stool Scale
  The seven types of stool are:
  Type 1: Separate hard lumps, like nuts (difficult to pass); Type 2: Sausage-shaped, but lumpy; Type 3: Like a sausage but with cracks on its surface; Type 4: Like a sausage or snake, smooth and soft (average stool); Type 5: Soft blobs with clear-cut edges; Type 6: Fluffy pieces with ragged edges, a mushy stool (diarrhea); Type 7: Watery, no solid pieces, entirely liquid (diarrhea)
Changes in the average eating time per meal | Day 7 compared to Day 0 and Day 28 compared to Day 0
  Changes in the average eating time per meal (minutes/meal)
Changes in the weight | Day 7 compared to Day 0 and Day 28 compared to Day 0
  Changes in the weight (kg)

SECONDARY OUTCOMES:
Changes in cytokines levels of blood samples | Day 28 compared to Day 0
  Changes in levels (pg/mL) in several cytokines, including tumor necrosis factor-α (TNF-α), interleukin-6 (IL-6), interleukin-10 (IL-10), interleukin-17 (IL-17), interleukin-23 (IL-23)
Changes in IgA levels in stool samples | Day 7 compared to Day 0 and Day 28 compared to Day 0
  Changes in levels (µg/mL) of pro-inflammatory IgA in stool samples
Changes in Intestinal microbiota | Day 28 compared to Day 0
  Changes in intestinal microbiota (bacterial phylum, family, genus, or species composition) in the stool samples of patients with constipation, anorexia, and slow weight gain before (Day 0) and after treatment (Day 28). Changes in intestinal microbiota: increase abundance of useful species and reduce abundance of harmful species
Changes ratio between the type of bacteria Gr (+), and Gr (-) | Day 7 compared to Day 0 and Day 28 compared to Day 0
  Changes in ratio between the type of bacteria Gr (+), and Gr (-) in the stool samples of patients with constipation, anorexia, and slow weight gain before (Day 0), middle (Day 7), and after treatment (Day 28)

CONTACTS AND LOCATIONS:
Overall Officials: Hanh TL Nguyen, PhD, Principal Investigator — National Institute of Nutrition (NIN), Ministry of Health, Vietnam
Locations (1):
- National Institute of Nutrition, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
Data or samples shared will be coded, with no PHI included. Approval of the request and execution of all applicable agreements (i.e., a material transfer agreement) are prerequisites to the sharing of data with the requesting party.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Data requests can be submitted 9 months after article publication and will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research. It will be provided following the review and approval of a study protocol, informed consent form (ICF), and clinical study report (CSR). For more information or to submit a request, please get in touch with clinicaltrial.probiotics@gmail.com

REFERENCES:
- [Background] Levy EI, Lemmens R, Vandenplas Y, Devreker T. Functional constipation in children: challenges and solutions. Pediatric Health Med Ther. 2017 Mar 9;8:19-27. doi: 10.2147/PHMT.S110940. eCollection 2017. PMID 29388621
- [Background] Chang CW, Chen MJ, Shih SC, Chang CW, Chiau JC, Lee HC, Lin YS, Lin WC, Wang HY. Bacillus coagulans (PROBACI) in treating constipation-dominant functional bowel disorders. Medicine (Baltimore). 2020 May;99(19):e20098. doi: 10.1097/MD.0000000000020098. PMID 32384482
- [Background] Dong M, Wu Y, Zhang M, Chen P, Zhang Z, Wang S. Effect of probiotics intake on constipation in children: an umbrella review. Front Nutr. 2023 Sep 1;10:1218909. doi: 10.3389/fnut.2023.1218909. eCollection 2023. PMID 37720380
- [Background] Freedman KE, Hill JL, Wei Y, Vazquez AR, Grubb DS, Trotter RE, Wrigley SD, Johnson SA, Foster MT, Weir TL. Examining the Gastrointestinal and Immunomodulatory Effects of the Novel Probiotic Bacillus subtilis DE111. Int J Mol Sci. 2021 Feb 28;22(5):2453. doi: 10.3390/ijms22052453. PMID 33671071
- [Background] Huang R, Hu J. Positive Effect of Probiotics on Constipation in Children: A Systematic Review and Meta-Analysis of Six Randomized Controlled Trials. Front Cell Infect Microbiol. 2017 Apr 28;7:153. doi: 10.3389/fcimb.2017.00153. eCollection 2017. PMID 28503492
- [Background] Bekkali NL, Bongers ME, Van den Berg MM, Liem O, Benninga MA. The role of a probiotics mixture in the treatment of childhood constipation: a pilot study. Nutr J. 2007 Aug 4;6:17. doi: 10.1186/1475-2891-6-17. PMID 17683583
- See also: UNICEF/WHO/The World Bank. 2021. Levels and trends in child malnutrition. World Health Organization. ISBN: 9789240025257 — https://www.who.int/publications/i/item/9789240025257